CLINICAL TRIAL: NCT00031993
Title: A Phase II Evaluation Of OSI-774 (NSC #718781) In The Treatment Of Persistent or Recurrent Squamous Cell Carcinoma Of The Cervix
Brief Title: Erlotinib in Treating Patients With Persistent or Recurrent Cancer of the Cervix
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02457; GOG-0227D; U10CA027469 (NIH); CDR0000069247 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Cervical Squamous Cell Carcinoma; Recurrent Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Erlotinib Hydrochloride

ARMS (1):
- Treatment (erlotinib hydrochloride) (Experimental): Patients receive oral erlotinib once daily for 4 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying erlotinib to see how well it works in treating patients with persistent or recurrent cancer of the cervix. Biological therapies such as erlotinib may interfere with the growth of tumor cells and slow the growth of the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the antitumor cytostatic activity of OSI-774 as measured by the probability of surviving progression-free for at least 6 months in patients with persistent or recurrent squamous cell carcinoma of the cervix.

II. To determine the nature and degree of toxicity of OSI-774 in this cohort of patients.

SECONDARY OBJECTIVES:

I. To determine the partial and complete response rates in patients with squamous cell carcinoma of the cervix receiving OSI-774.

II. To determine the duration of progression-free survival and overall survival within this patient population treated with OSI-774.

III. Assess the effects of prognostic factors: initial performance status and age.

TERTIARY OBJECTIVES:

I. To determine epidermal growth factor receptor (EGFR) and p110 truncated EGFR (p110 sEGFR) isoform expression levels in primary tumors, and from tumor samples obtained pretreatment and following four weeks of therapy to determine tumor response (or resistance) to OSI-774 inhibition of the EGFR tyrosine kinase.

II. To correlate EGFR and p110sEGFR expression levels with either MAPK or AKT phosphorylation status in the same tissue samples obtained pretreatment and following four weeks of drug treatment to determine downstream effects with response to OSI-774 inhibition of EGFR.

III. To determine whether pretreatment serum p110 sEGFR concentrations are a useful prognostic indicator and whether altered and/or sEGFR concentrations are useful indicators of therapeutic responsiveness, time to progression, and overall survival in cervical carcinoma patients.

OUTLINE: This is a multicenter study.

Patients receive oral erlotinib once daily for 4 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma (SCC) of the cervix

  * Persistent or recurrent progressive disease
  * At least 1 prior systemic chemotherapy regimen for management of advanced, metastatic, or recurrent SCC of the cervix is required

    * Chemotherapy administered as a radiosensitizer in conjunction with radiotherapy does not count as a systemic chemotherapy regimen
* At least 1 unidimensionally measurable target lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Lesions within a previously irradiated field are considered nontarget lesions unless disease progression or persistence is confirmed ≥ 90 days after completion of radiotherapy
* Tumor accessible for repeat needle biopsy
* Ineligible for a higher priority Gynecologic Oncology Group (GOG) protocol (any active GOG phase III protocol for the same patient population)
* Performance status - GOG 0-2 (for patients who have received only 1 prior regimen)
* Performance status - GOG 0-1 (for patients who have received 2 prior regimens)
* Platelet count at least 100,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Bilirubin no greater than upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No abnormalities of the cornea (e.g., dry eye syndrome or Sjogren's syndrome)
* No congenital abnormalities (e.g., Fuch's dystrophy)
* No abnormal slit-lamp examination using a vital dye (e.g., fluorescein or Bengal-Rose)
* No abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No uncontrolled concurrent illness
* No ongoing or active infection requiring IV antibiotics
* No psychiatric illness or social situation that would preclude study compliance
* No grade 2 or greater sensory or motor neuropathy
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to erlotinib
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* At least 3 weeks since prior immunologic therapy for SCC of the cervix
* One additional prior cytotoxic chemotherapy regimen for recurrent or persistent disease allowed
* At least 3 weeks since prior chemotherapy for SCC of the cervix and recovered
* No prior non-cytotoxic chemotherapy for recurrent or persistent disease
* At least 3 weeks since prior hormonal therapy for SCC of the cervix
* At least 3 weeks since prior radiotherapy for SCC of the cervix and recovered
* Recovered from recent prior surgery
* At least 3 weeks since other prior therapy for SCC of the cervix
* No prior epidermal growth factor receptor-targeting therapies
* No prior anticancer treatment that would preclude study participation
* No other concurrent investigational or commercial agents or therapies for SCC of the cervix

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2002-03; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | At 6 months
Frequency and severity of adverse effects as measured by NCI CTC version 3.0 | Up to 5 years

SECONDARY OUTCOMES:
Duration of overall survival | Up to 5 years
Duration of progression-free survival | Up to 5 years
Frequency of clinical response (complete and partial) | Up to 5 years
Prognostic factors including initial performance status and age | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schilder, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States